CLINICAL TRIAL: NCT03056937
Title: Effects of Bariatric Surgery on Inspiratory Metaboreflex in Metabolically Healthy Obese and Obese Subjects With Metabolic Syndrome
Brief Title: Effects of Bariatric Surgery on Inspiratory Metaboreflex in Obese Subjects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cruz Alta (Other)
Responsible Party: Sponsor
Other Study IDs: CAAE: 51573315.7.0000.5322
Record Dates: First submitted 2017-02-14; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese with metabolic syndrome: bariatric surgery
  Interventions: Other: Bariatric surgery
- Obese without metabolic syndrome: bariatric surgery
  Interventions: Other: Bariatric surgery
- Healthy: Control
  Interventions: Other: Control

INTERVENTIONS:
Other: Bariatric surgery — evaluations pre and post bariatric surgery.
  Groups: Obese with metabolic syndrome; Obese without metabolic syndrome
Other: Control — without intervention, it will be performed only evaluations
  Groups: Healthy

SUMMARY:
The hypothesis of this study is that reductions in body weight could improve inspiratory muscle function attenuating the inspiratory metaboreflex in metabolically healthy obese individuals and obese individuals with metabolic syndrome.

DETAILED DESCRIPTION:
Introduction: Peripheral metaboreflex activation appears to be exacerbated in obese individuals with metabolic syndrome. Interestingly, bariatric surgery attenuates the peripheral metaboreflex. Obese individuals have impaired inspiratory muscle function, which can be reversed by the reduction in body weight. Therefore, bariatric surgery could attenuate inspiratory metaboreflex in metabolically healthy obese individuals and obese individuals with metabolic syndrome. Objectives: To investigate the effects of bariatric surgery on inspiratory metaboreflex in metabolically healthy obese individuals and in obese patients with metabolic syndrome. Patients and Methods: A sample comprising of 15 obese subjects with metabolic syndrome, 15 obese subjects without metabolic syndrome and 15 healthy nonobese individuals. These subjects will be submitted to pulmonary function, respiratory muscle strength, inspiratory muscle resistance, exercise tolerance, quality of life, autonomic cardiovascular control and the inspiratory metaboreflex evaluation. The evaluations performed in obese patients with and without metabolic syndrome pre-surgery will be repeated 6 months after bariatric surgery.

ELIGIBILITY:
Obese with Metabolic Syndrome

Inclusion Criteria:

* Body mass index (BMI)> 35 kg / m²
* Diagnosis of metabolic syndrome

Exclusion Criteria:

* Acute health problems in the last month (viral or bacterial infections, accidents, allergic reactions)
* Diseases of the nervous system or conditions that affect the understanding or participation in the study
* Pregnancy
* Type I diabetes mellitus
* Arterial hypertension
* Dyslipidemias
* Coronary artery disease
* Left ventricular dysfunction
* Any condition interfering with locomotion
* Bronchial asthma
* Chronic obstructive pulmonary disease
* Chronic neuropathies
* Use of drugs such as corticosteroids or bronchodilators
* Smokers.

Obese without Metabolic Syndrome

Inclusion Criteria:

* Body mass index (BMI)> 35 kg / m²

Exclusion Criteria:

* Metabolic Syndrome
* Acute health problems in the last month (viral or bacterial infections, accidents, allergic reactions)
* Diseases of the nervous system or conditions that affect the understanding or participation in the study
* Pregnancy
* Type I diabetes mellitus
* Arterial hypertension
* Dyslipidemias
* Coronary artery disease
* Left ventricular dysfunction
* Any condition interfering with locomotion
* Bronchial asthma
* Chronic obstructive pulmonary disease
* Chronic neuropathies
* Use of drugs such as corticosteroids or bronchodilators
* Smokers.

Healthy nonobese subjects

Inclusion Criteria:

* BMI <25 kg / m²

Exclusion Criteria:

* Non-smokers
* Any diagnosed disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Obese subjects with metabolic syndrome, obese without metabolic syndrome and healthy nonobese subjects
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Inspiratory metaboreflex | 6 monhs
  It will be induced through a linear inspiratory resistance of 60% of maximal inspiratory pressure

SECONDARY OUTCOMES:
Pulmonary function | 6 months
  It will be assessed by spirometry
Respiratory muscle strength | 6 months
  It will be determined by manovacuometry.
Inspiratory muscle resistance | 6 months
  It will be evaluated through a protocol with progressive increase in inspiratory resistance.
Autonomic cardiovascular control | 6 months
  It will be determined by spectral analysis
Exercise tolerance | 6 months
  It will be determined by the 6-minute walk test.
Quality of life | 6 months
  It will be determined through the SF36 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Carine C Callegaro, PhD, Principal Investigator — University of Cruz Alta
Locations (1):
- University of Cruz Alta, Cruz Alta, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No